CLINICAL TRIAL: NCT05464251
Title: Prospective Analysis of Spinal Epidural Abscess Associated Outcomes at the University of Kentucky
Brief Title: Prospective Analysis of Spinal Epidural Abscess
Acronym: SEA
Status: Recruiting | Type: Observational
Sponsor: University of Kentucky (Other)
Responsible Party: Principal Investigator, Francis Farhadi, Associate Professor, University of Kentucky
Other Study IDs: 78749
Record Dates: First submitted 2022-06-28; First posted 2022-07-19 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Spinal Epidural Abscess
MeSH Terms: conditions — Epidural Abscess

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subjects with spinal epidural abscess with a history of drug abuse
  Interventions: Other: Prospective chart review of subjects diagnosed with spinal epidural abscess
- Subjects with spinal epidural abscess with no history of drug abuse
  Interventions: Other: Prospective chart review of subjects diagnosed with spinal epidural abscess

INTERVENTIONS:
Other: Prospective chart review of subjects diagnosed with spinal epidural abscess — Collection and assessment of available clinical, pathological, radiological, and socioeconomic data on subjects presenting with spinal epidural abscess. Standard of care treatment and outcomes for each group will be analyzed.

SUMMARY:
This is a prospective study involving all patients treated at the University of Kentucky for spinal epidural abscess over a 2-year period. Based on ongoing referrals of patients with SEA, we expect that 200 patients will be enrolled during this time window. We propose to study all available clinical, pathological, radiological, and socioeconomic data of patients diagnosed with a spinal infection with or without a history of drug abuse over this study period. All patients' charts will be prospectively reviewed starting at the time of presentation for a period of 1 year.

ELIGIBILITY:
Inclusion Criteria:

* All patient with ICD codes for pyogenic vertebral osteomyelitis, discitis, and spinal epidural abscess will be reviewed for inclusion.

Exclusion Criteria:

* Patients unwilling or unable to attend follow up appointments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include all patients, over the age of 18, who will undergo treatment for spinal epidural abscess infections at the University of Kentucky during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-07-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Correlation between employment status and infection reoccurrence. | 1 year
  Determine the statistical correlation between employment status and infection reoccurrence within 1 year of diagnosis.
Correlation between income and infection reoccurrence. | 1 year
  Determine the statistical correlation between income and infection reoccurrence within 1 year of diagnosis.
Correlation between insurer and infection reoccurrence. | 1 year
  Determine the statistical correlation between insurer (private, Medicare/Medicade and uninsured) and infection reoccurrence within 1 year of diagnosis.
Correlation between living situation and infection reoccurrence. | 1 year
  Determine the statistical correlation between living situation (owns, rents, or homeless) and infection reoccurrence within 1 year of diagnosis.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Undecided